CLINICAL TRIAL: NCT01366170
Title: Expression of T Immunoregulatory Proteins in ALK+ Anaplastic Large Cell Lymphoma (ALCL)
Brief Title: Biomarker Expression in Samples From Young Patients With Anaplastic Large Cell Lymphoma
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANHL11B1; COG-ANHL11B1 (Other: Children's Oncology Group); NCI-2011-02860 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ANHL11B1 (Other: Children's Oncology Group)
Record Dates: First submitted 2011-06-02; First posted 2011-06-03 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Lymphoma
Keywords: childhood anaplastic large cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Large-Cell, Anaplastic | interventions — Microarray Analysis; Blotting, Western; Flow Cytometry; Immunohistochemistry; Mass Spectrometry

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: microarray analysis
Genetic: protein expression analysis
Genetic: western blotting
Other: flow cytometry
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: mass spectrometry

SUMMARY:
RATIONALE: Studying samples of tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer. it may also help doctors predict how patients will respond to treatment.

PURPOSE: This research trial studies biomarker expression in tissue samples from young patients with anaplastic large cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the expression of immunoregulatory proteins including CD4, FOXP3 and CD276 in anaplastic large cell lymphoma (ALCL).
* To correlate the expression of these proteins with the levels of anaplastic lymphoma kinase (ALK) autoantibodies in patient of ANHL0131.

OUTLINE: Archived tissue microarray samples are analyzed by mass spectrometry and validated by Western blotting, flow cytometry, and IHC.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of anaplastic large cell lymphoma
* Tissue microarray samples available from the Cooperative Human Tissue Network (CHTN)

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Max Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Diagnosis of anaplastic large cell lymphoma.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Estimated)
Dates: Start 2011-05; Primary Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Expression of immunoregulatory proteins including CD4, FOXP3 and CD276 in ALCL
Correlation of CD4, FOXP3, and CD276 with ALK autoantibody response in patients enrolled in ANHL0131

CONTACTS AND LOCATIONS:
Overall Officials: Megan S. Lim, MD, PhD, Principal Investigator — C.S. Mott Children's Hospital at University of Michigan Medical Center